CLINICAL TRIAL: NCT02913768
Title: Reduction in Spinal-induced Hypotension With Ondansetron in Parturients Undergoing Caesarean Section: A Double-blind Randomised, Placebo-controlled Study
Brief Title: Reduction in Spinal-induced Hypotension With Ondansetron in Parturients Undergoing Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, lecturer of anesthesia and ICU, Assiut University,Assiut, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ondansetron for CS
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Ondansetron (Active Comparator): Intravenous Ondansetron 4 mg diluted in 10 mL of normal saline over 1 min, 5 min before spinal anaesthesia
  Interventions: Drug: Ondansetron
- control (Placebo Comparator): Normal Saline 10 mL over 1 min, 5 min before spinal anaesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ondansetron
  Arms: Ondansetron
Drug: Normal saline
  Arms: control

SUMMARY:
Subarachnoid block is the preferred method of anaesthesia for caesarean section, but is associated with hypotension and bradycardia, which may be deleterious to both parturient and baby. Animal studies suggest that in the presence of decreased blood volume, 5-HT may be an important factor inducing the Bezold Jarisch reflex via 5-HT3 receptors located in intracardiac vagal nerve endings. In this study, the investigators evaluated the effect of ondansetron, as a 5-HT3 receptor antagonist, on the haemodynamic response following subarachnoid block in parturients undergoing elective caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an elective lower segment caesarean section.

Exclusion Criteria:

* Patients with contraindications to subarachnoid block (patient refusal, unstable haemodynamics, coagulation abnormality),
* History of hypersensitivity to ondansetron or local anaesthetic agents,
* Hypertensive disorders of pregnancy,
* Cardiovascular insufficiency,
* Receiving selective serotonin reuptake inhibitors or migraine medications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Hypotension | intraoperative
  Systolic BP <90 mmHg or Diastolic BP <60 mmHg

SECONDARY OUTCOMES:
Bradycardia | intraoperative
  HR <50 beats/min

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt